CLINICAL TRIAL: NCT01747785
Title: Myocardial Performance at Rest and During Exercise in Heart Failure With Preserved Ejection Fraction: Speckle Tracking Echocardiography - One Piece of the Puzzle.
Brief Title: Myocardial Performance at Rest and During Exercise in Heart Failure With Preserved Ejection Fraction
Acronym: X-HF-SPECKLE
Status: Terminated | Type: Observational
Why Stopped: Study stopped for administrative reasons.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hector R. Villarraga, M.D., PI, Mayo Clinic
Other Study IDs: 12-005553
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure
Keywords: Heart failure; HFpEF; Dyspnea; Fatigue; Shortness of Breath; exercise; strain; myocardial deformation; cardiac rehabilitation; cardiac hemodynamics
MeSH Terms: conditions — Heart Failure; Dyspnea; Fatigue; Motor Activity; Sprains and Strains | interventions — Cardiac Rehabilitation; Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy controls: Individuals without history of cardiovascular disease and at least 18 years of age will take a baseline (at rest) cardiopulmonary exercise test (CPX) and have a cardiac echocardiogram to measure myocardial deformation. CPX and echocardiograms will be repeated during exercise sessions at 3 visits over a 12 week period.
  Interventions: Other: Myocardial deformation imaging; Other: Cardiopulmonary exercise test
- Patients at risk of heart failure: Individuals at risk of heart failure and a preserved ejection fraction of at least 50% will take a baseline (at rest) cardiopulmonary exercise test (CPX) and have a baseline cardiac echocardiogram to measure myocardial deformation. CPX and echocardiograms will be repeated during exercise sessions at 6 visits over a 12 week period. A cardiac rehabilitation exercise program will also occur over 12 weeks.
  Interventions: Other: Cardiac rehabilitation; Other: Myocardial deformation imaging; Other: Cardiopulmonary exercise test

INTERVENTIONS:
Other: Cardiac rehabilitation — Aerobic cardiac exercise training will be provided over the 12 week study duration.
  Groups: Patients at risk of heart failure
Other: Myocardial deformation imaging — A 2D Doppler echocardiograph (image) of the heart will be captured during a single heart beat taken at rest and during cardiopulmonary exercise tests to measure left and right ventricular segmental systolic and diastolic strain measurements.
Other: Cardiopulmonary exercise test — The cardiopulmonary exercise test consists of cycling exercise of mild and moderate intensity on an upright cycle ergometer on a tilting table (to facilitate imaging) for 6-10 minute periods within a one hour session.

SUMMARY:
This study is being done to study how well the heart contracts and relaxes during exercise. In addition to traditional measures of heart function, we will use a new computer program that may improve understanding of why people feel shortness of breath or fatigue.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction is not well understood, although account for nearly half of all heart failure cases. This study aims to collect data about systolic (contracting portion of a heart beat) and diastolic (relaxing portion of a heart beat) dysfunction at rest and during exercise. Participants with normal cardiac function will serve as a control group and compared to participants who are at risk of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* able to exercise on a bicycle

Exclusion Criteria:

* heart arrhythmias,
* severe chronic obstructive pulmonary disease,
* congenital heart abnormalities,
* infiltrative or hypertrophic cardiomyopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in mean cardiac reserve as measured by strain rate | Baseline, 12 weeks
  Myocardial deformation imaging (e.g. strain, strain rate, torsion) requires clear 2-dimensional echocardiography images that will be obtain at rest and during mild and moderate intensity exercise. Images will be captured during 6-10 minute bouts of exercise on a tilting exercise table. Comparisons will be made on resting and exercise values between groups. Our hypothesis is that strain rate will not increase in patients at risk of heart failure demonstrating lack of cardiovascular reserve.

SECONDARY OUTCOMES:
Change in mean cardiac stroke volume | Baseline, 12 weeks
  Stroke volume is the volume of blood (in milliliters) ejected during each heart contraction, It is measured by combined Doppler and 2-dimensional echocardiography. A surrogate measure of stroke volume (oxygen-pulse) can also be obtained during cardiopulmonary exercise testing by dividing the measured oxygen consumption by the heart rate. Our hypothesis is that stroke volume will plateau early after exercise onset in patients at risk of heart failure and this plateau will correlate with a reduction in strain rate.

CONTACTS AND LOCATIONS:
Overall Officials: Hector Villarraga, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System - Franciscan Healthcare, La Crosse, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No